CLINICAL TRIAL: NCT05683093
Title: Cardiovascular Longitudinal the Avon Longitudinal Study of Parents and Children (ALSPAC) Research Investigations Following Hypertensive Pregnancy in Young Adulthood
Brief Title: Cardiovascular Longitudinal ALSPAC Research Investigations Following Hypertensive Pregnancy in Young Adulthood
Acronym: CLARITY
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: 22/WA/0227
Record Dates: First submitted 2022-11-07; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Young Adult; Hypertension in Pregnancy; Hypertension; Cardiovascular Diseases; Cerebrovascular Diseases; Vascular Diseases
Keywords: Young Adult; Birth History; Hypertension in Pregnancy; Cardiovascular Risk; Exercise Capacity
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Cardiovascular Diseases; Cerebrovascular Disorders; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: History of being born to hypertensive or normal pregnancy — CLARITY is an observational study whereby participants will attend one 4-hr visit the Division of Cardiovascular Medicine, University of Oxford at the John Radcliffe Hospital in Oxford, with the option to split the study visit over two days for convenience.
  Participants will be invited by the ALSPAC study team to attend a study visit in Oxford where the investigators will use MRI and other imaging modalities to study the brain, heart, liver, kidneys, and vasculature using standardised protocols. A dataset including information from previous follow-up of these cohorts and the detailed pregnancy data available within ALSPAC will be generated by the study team in Bristol and integrated with available data from the Oxford cohorts.

SUMMARY:
The purpose of this study is to understand more about why young people who were born to a hypertensive pregnancy may have increased risk of high blood pressure and are often at increased risk of heart and blood vessel disease later in life.

DETAILED DESCRIPTION:
Women who develop blood pressure problems during pregnancy are more likely to have high blood pressure (hypertension) in later life as well as heart attacks or strokes. The children born to the pregnancy also tend to have higher blood pressure and are often at increased risk of heart and blood vessel disease later in life. Previous work has shown that children born to pregnancies where the mother has high blood pressure have changes in their blood vessels, heart and brain that can be measured long before they develop high blood pressure or other clinical symptoms. By understanding the pattern of changes cross multiple parts of the body, over a lifetime, the investigators can identify how advanced the underlying disease is for an individual and how their disease is likely to develop over the next few years.

The aim of this study is to understand the heart and blood vessel changes of people born to a hypertensive pregnancy once they are in their 20s and 30s. The investigators then hope to use this information to develop new ways to prevent early onset heart and blood vessel disease in these people.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or female, aged 30 to 40 years at time of enrolment
* Participant previously took part in the ALSPAC study
* Able (in the investigator's opinion) and willing to comply with all study requirements
* Adequate understanding of verbal and written English

Exclusion Criteria:

* Pregnant or lactating when they are due to attend for study visit 1
* Less than six months postpartum
* Planning to donate blood within two weeks prior to study visit 1
* Any significant disease or disorder which, in the opinion of the investigator, might influence the participant's ability to participate in the study
* Evidence of congenital heart disease or significant chronic disease relevant to cardiovascular or metabolic status

For exclusion of MRI component only:

* Unsuitable for MRI based on participant screening; the participant may still be included in other parts of the study

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Of the 200 young adults followed up from the ALSPAC study, 100 will have been born to a hypertensive pregnancy and 100 following an uncomplicated pregnancy. At time of follow-up, they will be 30 to 40 years of age. At the 25-year follow-up in Bristol, there were 610 individuals born to hypertensive pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac right ventricular mass | 30-40 years of old
  Magnetic resonance imaging (MRI) assessment of cardiac right ventricular mass indexed to body surface area (in g and g/m^2)

SECONDARY OUTCOMES:
Cardiac left ventricular mass | 30-40 years of old
  MRI assessment of cardiac left ventricular mass indexed to body surface area (in g and g/m^2)
Cardiac right ventricular end-diastolic volume | 30-40 years of old
  MRI assessment of cardiac right ventricular end-diastolic volume indexed to body surface area (in ml and ml/m^2)
Cardiac right ventricular stroke volume | 30-40 years of old
  MRI assessment of cardiac right ventricular stroke volume indexed to body surface area (in ml and ml/m^2)
Cardiac left ventricular end-diastolic volume | 30-40 years of old
  MRI assessment of cardiac left ventricular end-diastolic volume indexed to body surface area (in ml and ml/m^2)
Cardiac left ventricular stroke volume | 30-40 years of old
  MRI assessment of cardiac left ventricular stroke volume indexed to body surface area (in ml and ml/m^2)
Cardiac right ventricular systolic function | 30-40 years of old
  Echocardiography and MRI assessment of right ventricular systolic function: tricuspid annular plane systolic excursion (in cm) and right ventricular ejection fraction measured by cardiac MRI (in %)
Cardiac left ventricular systolic function | 30-40 years of old
  Echocardiography and MRI assessment of left ventricular systolic function: left ventricular ejection fraction (in %)
Cardiac right ventricular diastolic function | 30-40 years of old
  Echocardiography assessment of right ventricular (RV) diastolic function: RV Doppler early/late diastolic tricuspid inflow velocity ratio (E/A)
Cardiac left ventricular diastolic function | 30-40 years of old
  Echocardiography assessment of left ventricular (LV) diastolic function: LV Doppler early/late diastolic mitral inflow velocity ratio (E/A) and LV early Doppler inflow velocity/peak early diastolic tissue velocity ratio (E/e')
Morphology of the right ventricles | 30-40 years of old
  MRI assessment of the right ventricles morphology using cardiac statistical atlas and principal component analysis
Morphology of the left ventricles | 30-40 years of old
  MRI assessment of the left ventricles morphology using cardiac statistical atlas and principal component analysis
Aortic compliance | 30-40 years of old
  Aortic distensibility by MRI (in 10^-3 mmHg^-1) and aortic/central blood pressure by cuff measurement (in mmHg)
Intra-hepatic lipid content, steatohepatitis and hepatic fibrosis | 30-40 years of old
  MRI assessment of the liver to quantify proton density fat fraction (in %) and fibro-inflammatory status from iron-corrected T1 (cT1 in ms)
Renal function | 30-40 years of old
  MRI assessment of fibro-inflammatory status from T1 (in ms) and surrogate measure of blood perfusion from T2* (in ms) and volumes (in ml and ml/m^2)
Oxygen uptake across sub-maximal and peak exercise | 30-40 years of old
  Cardiopulmonary exercise test to measure oxygen uptake (VO2 in ml/kg/min)
Carbon dioxide exchange kinetics across sub-maximal and peak exercise | 30-40 years of old
  Cardiopulmonary exercise test to measure respiratory exchange ratio (RER calculated as carbon dioxide production divided by oxygen consumption)
Retinal arteriolar structure | 30-40 years of old
  Central retinal arteriolar equivalent (CRAE in μm) measured using retinal imaging
Retinal venular structure | 30-40 years of old
  Central retinal venular equivalent (CRVE in μm) measured using retinal imaging
Retinal arteriolar-to-venular diameter ratio (AVR) | 30-40 years of old
  The ratio of average retinal arteriolar diameter (CRAE in μm) and average retinal venous diameter (CRVE in μm) measured using retinal imaging
Ear microvascular structure | 30-40 years of old
  Superior crus of anti-helix earlobe vascular caliber (in μm) measured using ear vascular imaging
Lung function | 30-40 years of old
  The forced expiratory volume in one second (FEV1 in L), forced vital capacity (FVC in L), and the ratio of FEV1 to FVC (FEV1/FVC) measured using spirometry
Objective measure of physical activity | 30-40 years of old
  The amount of moderate to vigorous physical activity (in h/week) and vigorous physical activity (in h/week) measured using wrist worn accelerometer
Total white matter volume | 30-40 years of old
  Total white matter volumes (in mm3) assessed on T1-weighted sequence of brain MRI
Total grey matter volume | 30-40 years of old
  Total grey matter volumes (in mm3) assessed on T1-weighted sequence of brain MRI
Subcortical brain volume of thalamus | 30-40 years of old
  Subcortical brain volume of thalamus (in mm3) assessed on T1-weighted sequence of brain MRI
Subcortical brain volume of hippocampus | 30-40 years of old
  Subcortical brain volume of hippocampus (in mm3) assessed on T1-weighted sequence of brain MRI
White matter hyperintensities volume | 30-40 years of old
  Total volume of white matter hyperintensities (in mm3) assessed on T2-weighted sequence of brain MRI
White matter hyperintensities count | 30-40 years of old
  The number of white matter hyperintensities on T2-weighted sequence of brain MRI
Cerebral vessel lumen diameter | 30-40 years of old
  Cerebral vessel lumen diameter (in μm) assessed on the time-of-flight sequence of brain MRI
Cerebral vessel density | 30-40 years of old
  Cerebral vessel density (in mm3) assessed on the time-of-flight sequence of brain MRI
Cerebral vessel tortuosity | 30-40 years of old
  The ratio of cerebral vessel tortuosity assessed on the time-of-flight sequence of brain MRI
Whole brain grey matter perfusion or cerebral blood flow (CBF) | 30-40 years of old
  Whole brain grey matter perfusion/CBF (in ml/100g/min) assessed on arterial spin labelling of brain MRI
Arterial cerebral blood volume fraction | 30-40 years of old
  Arterial cerebral blood volume fraction (in %) assessed on arterial spin labelling of brain MRI
Circulating vascular endothelial growth factor A (VEGF-A) as an angiogenic marker | 30-40 years of old
  The level of VEGF-A (in pg/mL) measured from plasma blood samples
Circulating soluble endoglin (sENG) as an angiogenic marker | 30-40 years of old
  The level of sENG (in ng/mL) measured from plasma blood samples
Circulating soluble fms-like tyrosine kinase-1 (sFlt-1) as an antiangiogenic marker | 30-40 years of old
  The level of sFlt-1 (in pg/mL) measured from plasma blood samples
Circulating total cholesterol as a metabolic marker | 30-40 years of old
  The level of total cholesterol (in mmol/L) measured from serum blood samples
Circulating high-density lipoprotein as a metabolic marker | 30-40 years of old
  The level of HDL (in mmol/L) measured from serum blood samples
Circulating low-density lipoprotein as a metabolic marker | 30-40 years of old
  The level of LDL (in mmol/L) measured from serum blood samples
Circulating triglycerides as a metabolic marker | 30-40 years of old
  The level of triglycerides (in mmol/L) measured from serum blood samples
Circulating fasting glucose concentration as a metabolic marker | 30-40 years of old
  The level of fasting glucose (in mmol/L) measured from whole blood samples
Circulating fasting insulin concentration as a metabolic marker | 30-40 years of old
  The level of fasting insulin (in pmol/L) measured from serum blood samples
Insulin resistance index (HOMA-IR) as a metabolic marker | 30-40 years of old
  The index calculated as fasting glucose (in mmol/L) x fasting insulin (in μIU/mL) ÷ 22.5
Circulating C-reactive protein (CRP) as an inflammatory marker | 30-40 years of old
  The level of CRP (in mmol/L) measured from serum blood samples
Circulating soluble intercellular adhesion molecule-1 (sICAM-1) as an inflammatory marker | 30-40 years of old
  The level of sICAM-1 (in ng/mL) measured from serum blood samples
Circulating soluble vascular cell adhesion molecule-1 (sVCAM-1) as an inflammatory marker | 30-40 years of old
  The level of sVCAM-1 (in ng/mL) measured from serum blood samples
Body weight | 30-40 years of old
  Body weight measured in kg
Body height | 30-40 years of old
  Body height measured in m
Body mass index | 30-40 years of old
  Body weight divided by the square of height (in kg/m2)
Mid-arm circumference | 30-40 years of old
  Mid-arm circumference measured in cm
Waist-to-hip ratio | 30-40 years of old
  The ratio of waist circumference (in cm) to hip circumference (in cm)
Systolic blood pressure | 30-40 years of old
  Resting brachial blood pressure measurement (in mmHg)
Diastolic blood pressure | 30-40 years of old
  Resting brachial blood pressure measurement (in mmHg)
Mean arterial pressure | 30-40 years of old
  The average arterial pressure from resting brachial blood pressure measurement (in mmHg)
Pulse pressure | 30-40 years of old
  The difference between systolic and diastolic blood pressure (in mmHg)
Heart rate | 30-40 years of old
  The frequency of the heart contractions per minute (in beats per minute or bpm)
Smoking status | 30-40 years of old
  The number and percentage of current smokers
Alcohol consumption | 30-40 years of old
  Weekly alcoholic unit intake (in units per week)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Lewandowski, Principal Investigator — Cardiovascular Clinical Research Facility
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No